CLINICAL TRIAL: NCT04932707
Title: Effect of Adding Suboccipital Muscle Release Versus Neurodynamic Mobilization to Passive Hamstring Stretch in Subjects With Short Hamstring Syndrome.
Brief Title: Stretching Exercises on Hamstring Flexibility.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Olfat Ibrahim Ali, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hamstring muscle shortening
Record Dates: First submitted 2021-06-12; First posted 2021-06-21 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Hamstring Muscle; Flexibility
Keywords: hamstring; Stretch; Sub-occipital inhibition; Neuro-dynamic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group 1 (Experimental): sub-occipital muscle inhibition.
  Interventions: Other: sub-occipital muscle inhibition technique; Other: control (passive stretch exercises)
- Study group 2 (Experimental): Received neurodynamic mobilization.
  Interventions: Other: Neurodynamic mobilization; Other: control (passive stretch exercises)
- control group (Active Comparator): Received passive stretch of the hamstring muscle.
  Interventions: Other: control (passive stretch exercises)

INTERVENTIONS:
Other: sub-occipital muscle inhibition technique — this technique will be conducted from a supine lying position. The therapist stretches the suboccipital, placing the hands beneath the patient's head applying pressure up and backward, pressure was maintained till tissue relaxation occurred flexes the head of the patient to get the chin to the manibiurim sternm.
  Arms: Study group 1
Other: Neurodynamic mobilization — Patient in a comfortable short sitting position at the edge of the bed with the trunk in an military straight position then ask the patient to slump; flex her neck and street the knee joint in complete extension the at the end of the procedure do active dorsiflexion at the tested foot.
  Arms: Study group 2
Other: control (passive stretch exercises) — The patient in a comfortable supine lying position, the patient was asked to flex his hip joint with complete knee extension and ankle in neutral position. The therapist stretches the hamstring of the dominant side

SUMMARY:
The hamstrings muscles are examples of muscle groups that have a tendency to shorten.

Limited flexibility has been shown to predispose a person to several musculoskeletal overuse injuries and significantly affect a person's function.

DETAILED DESCRIPTION:
The objective of this study will be to compare the effect of three different methods of stretching techniques on the flexibility of hamstring muscle in subjects with short hamstring syndrome.

HYPOTHESES:

There will be no difference between sub-occipital muscle inhibition technique, neuro-dynamic slump stretch, or passive hamstring stretch on hamstring flexibility in subjects with short hamstring syndrome.

RESEARCH QUESTION:

Is there is any difference between suboccipital muscle inhibition technique, neurodynamic slump stretch, or passive hamstring stretch on hamstring flexibility in patients with short hamstring syndrome?

ELIGIBILITY:
Inclusion Criteria:

* undergraduate female students
* body mass index 18-25 kg/cm square.
* All subjects will be free from injury or disease expected to affect hamstring length or ability to perform the exercises.

Exclusion Criteria:

* Hamstring injury within the past year.
* Verbal report of performing regular lower extremity.
* Current Muscle stretching exercises.
* History of neck trauma (whiplash).
* History of recent fracture in any part of the body.
* History of neurological or orthopedic disorders
* Diagnosis of a herniated disk
* Low back pain in the last 6 months

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2023-07-16 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
knee extension angle test | Immediately after the procedure
  Measure the knee extension knee joint from a supine lying position with hip and knee joints flexed to 90 degree.
knee extension angle test | 4 weeks
  Measure the knee extension knee joint from a supine lying position with hip and knee joints flexed to 90 degree.

SECONDARY OUTCOMES:
Straight leg raising test | Immediately after the procedure
  Patient asked to raise her leg with extended knee and measure the hip joint jt flexion angle
Straight leg raising test | 4 weeks
  Patient asked to raise her leg with extended knee and measure the hip joint jt flexion angle
Forward flexion test | Immediately after the procedure
  subjects were asked to flex her trunk with his hands facing forward, maintaining the knee in extended position and measure the distance between hand ground
Forward flexion test | 4 weeks
  subjects were asked to flex her trunk with his hands facing forward, maintaining the knee in extended position and measure the distance between hand ground

CONTACTS AND LOCATIONS:
Overall Officials: Olfat I Ali, PhD, Principal Investigator — Cairo University
Locations (1):
- Olfat Ibrahim Ali, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Sharing will be possible after the publication of the study
Supporting Information: Study Protocol
Time Frame: After study publication
Access Criteria: Contact: Olfat Ibrahim Ali, email address: olfat_ib@yahoo.com, olfat_ib@cu.edu.eg